CLINICAL TRIAL: NCT05143775
Title: Strategic Intervention on Preserving Language Function During Awake Craniotomy for Glioma Resection
Brief Title: Strategic Intervention on Preserving Language Function During Awake Craniotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY 2020-099-01
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Glioma
Keywords: functional preservation; awake craniotomy; language impairment
MeSH Terms: conditions — Glioma; Language Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new surgical plan group (Experimental): The investigators use a monopolar stimulator to determine and retain the tumor margin within 5mm in the sensitive area which is posterior superior longitudinal fasciculus or posterior arcuate fasciculus.
  Interventions: Procedure: Awake craniotomy
- traditional surgical plan group (Active Comparator): The investigators use bipolar stimulator according to the current standard surgery plan. After the positive points are identified, those points would be retained to avoiding language function impairment after the tumor resection.
  Interventions: Procedure: Awake craniotomy

INTERVENTIONS:
Procedure: Awake craniotomy — Randomly select 30 participants to implement new surgical plan, which is using a monopolar stimulator to determine positive function sites and save tumors within 5 mm of the posterior superior longitudinal fasciculus/arcuate fasciculus

SUMMARY:
This study is designed to compare the language function after traditional or a new surgical plan during awake craniotomy for glioma resection.

DETAILED DESCRIPTION:
This study concentrates on patient who has type II language area glioma occupation. The investigators designed new surgical plan which is using monopolar stimulator to determine and retain the tumor margin within 5 mm from the posterior superior longitudinal fasciculus or posterior arcuate fasciculus. For the tradiitional surgical plan, the investigators use bipolar stimulator according to the current standard surgery plan. After they positive points are identified by stimulator, the positive points are retained to preserve the motor function while all the negative points of the tumor are resected. This study is to determine whether the new surgical plan is more suitable for type II language area glioma occupation.

ELIGIBILITY:
Inclusion Criteria:

1, patients with glioma near or on the language function area that have the necessity to undergo awake craniotomy and language function identification during tumor resection

Exclusion Criteria:

1. patients with incompleted monitoring procedures;
2. paitents without data of the pre-and postoperative resting state MRI, diffuison tensor image and functional MRI.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change of the language impairment rate | From date of the first tumor resection until the date of death from any cause, assessed up to 500 months.
  The ratio of language function recovery in patients with new surgical plan would higher than those receive traditional surgical plan. The main tool is to use Western Aphasia Battery (WAB) language evaluation form to record each patient's language ability in 4-7days after surgery and every other 3 months. The executive function and attention would also be evaluated by cognitive assessment (MoCA) and Mini-Mental State Exam (MMSE). Each patient's scores and reponse time would be used to compare the differences between two surgical plans.
Change of the survival rate | From date of the first tumor resection until the date of death from any cause, assessed up to 500 months.
  The new surgical plan preserves the language function to improve the quality of life, in order to influence the patient's length of life after surgery. Hence, the overall survival days of patients in two surgical plans would be compared by recording patients' date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Tao, Study Chair — Beijing Neurosurgical Institute
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The investigators don't plan to share individual participant data with other researchers

REFERENCES:
- [Background] Fang S, Liang Y, Li L, Wang L, Fan X, Wang Y, Jiang T. Tumor location-based classification of surgery-related language impairments in patients with glioma. J Neurooncol. 2021 Nov;155(2):143-152. doi: 10.1007/s11060-021-03858-9. Epub 2021 Oct 1. PMID 34599481